CLINICAL TRIAL: NCT04610242
Title: Prediction of Rituximab Hypersensitivity and Desensitization Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-Allergy-01
Record Dates: First submitted 2020-09-25; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-09

CONDITIONS: Drug Hypersensitivity Reaction
Keywords: Rituximab; Drug hypersensitivity reaction; Skin test; Desensitization
MeSH Terms: interventions — Skin Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients undergo diagnostic tests before the initial infusion of rituximab, including skin prick tests, intradermal tests, and challenge tests successively. If the skin test shows a positive result, the patient will receive desensitization procedure, and if the skin test is negative, the challenge test will be done, meaning normal infusion of rituximab according to manufacturer instructions. All the HSRs in the process of desensitization or normal infusion will be recorded. Peripheral blood will be drawn from all the subjects during their infusion to investigate the mechanism of HSRs to rituximab.
  Interventions: Diagnostic Test: skin test

INTERVENTIONS:
Diagnostic Test: skin test — For skin prick tests (SPT), rituximab solution of 1mg/ml was applied on the volar aspect of the forearm. For intradermal tests (IDT), 0.02 mL of a 1:100 dilution (0.1mg/ml) of full-strength solution (10mg/ml) was injected first. If the result was negative, a 1:10 dilution（1mg/ml）was then used.
  As to the desensitization protocol, three solutions with different concentrations are delivered in 12 consecutive steps, each step increasing the rate of drug administration by 2- to 2.5-fold. Solution 1 is a 100-fold dilution (0.01mg/ml) of the final target concentration, solution 2 is a 10-fold dilution (0.1mg/ml) of the final target concentration, and the concentration of solution 3 is the target concentration (1mg/ml). Each step takes 15 minutes until the target rate of 200ml/h is reached, and the final step is prolonged to complete the target dose. The whole procedure takes about 5.5 hours.
  Other Names: desensitization for patients with positive skin test results

SUMMARY:
This is a single-center prospective single arm study. The purpose of this study is to assess the usefulness of skin test as a diagnostic tool to predict the hypersensitivity to rituximab in Chinese population, evaluate the rate of hypersensitivity reactions (HSRs) after the application of active desensitization therapy in the case of a positive skin test result, and investigate the mechanism of HSRs to rituximab.

DETAILED DESCRIPTION:
Patients with B-cell lymphomas who need the administration of rituximab are recruited. They undergo skin tests with rituximab before the first infusion of this medicine. In the case of a positive skin test result, the patient will receive the desensitization procedure; if the result of skin test is negative, the challenge test will be administered. Drug challenge test consists in administering the desired full dose of rituximab according to manufacturer instructions. Challenge is considered positive when it shows an objective HSR. The patient with a positive challenge test will receive the desensitization procedure; while the patient with a negative challenge test will be given standard rituximab infusion in the subsequent chemotherapies.

Peripheral blood will be drawn from all the subjects during their initial infusion of rituximab. If the patient shows hypersensitive symptoms, the blood will be drawn one hour after the onset of reaction; while if the patient has no HSR in the whole infusion process, the blood will be drawn at the end of infusion and used as negative control. Levels of tryptase, specific immunoglobulin E to rituximab, IL-6, IL-8, and TNF-α in the serum will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B cell lymphoma confirmed through pathological biopsy
* Patients who need the treatment of rituximab and have not received rituximab before

Exclusion Criteria:

* Pregnant or lactating women
* Patients taking antihistamines in three days before the skin tests
* Long-term use of systemic corticosteroid
* Patients with skin lesions including infection, dermatitis, trauma or scar in both arms
* Patients with acute attack of asthma
* Patients with psoriasis
* Other conditions that the researchers consider inappropriate to participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of skin test | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  The sensitivity and specificity of skin test in the prediction of HSR to rituximab.

SECONDARY OUTCOMES:
Hypersensitivity reactions (HSRs) | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  The rate of HSRs in all the enrolled subjects with the application of active desensitization therapy in the case of a positive skin test result.
Tryptase | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  Level of serum tryptase
Specific immunoglobulin E to rituximab | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  Level of serum specific immunoglobulin E to rituximab
IL-6 | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  Level of serum IL-6
IL-8 | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  Level of serum IL-8
TNF-α | From date of signing the informed consent until the end of induction chemotherapy, up to 32 weeks
  Level of serum TNF-α

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No